CLINICAL TRIAL: NCT03973346
Title: Improving Population and Clinical Health With Integrated Services and Advanced Analytics
Brief Title: Impact of Social Risk Decision Support
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The implementation of the tool has been delayed due to technology governance issues and requests for changes in the end user design.
Sponsor: Indiana University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Joshua R. Vest, PhD, Associate Professor & Center Director, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: VEST-RWJF-PHASE2
Record Dates: First submitted 2019-05-28; First posted 2019-06-04 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Health Social Determinant
Keywords: risk prediction

STUDY DESIGN:
Intervention Model Description: Multiple observation, pre-post with a secondary data source comparison group design, and a difference-in-difference modeling approach.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Encounters at primary care clinics with the risk screening tool
  Interventions: Other: Risk screening tool exposure
- Comparison group (No Intervention): Propensity score matched comparison encounters

INTERVENTIONS:
Other: Risk screening tool exposure — Risk screening tool is available to providers
  Arms: Intervention group

SUMMARY:
The purpose of this study is to determine the impact of embedding a risk-stratification tool, designed to identify patient needs for services that address social determinant of health related needs, in a commercial electronic health record system (EHR).

DETAILED DESCRIPTION:
Social determinant of health related needs and social risk factors complicate care delivery and drive health and well-being. Social needs are common among undeserved patient populations, but health care providers are often not equipped to routinely identify and address patients in need.

Using a combination of health information exchange, electronic health record, and aggregate datasets the investigators developed predictive algorithms to identify patients a highest risk for a need for a referral to a social worker, dietitian, behavioral health, or other wraparound service provider. Risk scores are available to primary care providers in two ways within the electronic health record system (EHR): 1) a graphical summary of individual risk or 2) a line listing of all scheduled patients.

The investigators are introducing the risk-stratification tool in an urban safety-net primary care provider on a voluntary usage basis.

ELIGIBILITY:
Inclusion Criteria:

* Encounters among patients seeking primary care service at any of the 9 Eskenazi Health FQHC clinics in Indianapolis, IN from January 2017 to May 2020.
* The propensity score matched primary care encounters from non-Eskenazi facilities.

Exclusion Criteria:

* Emergency encounters or hospitalizations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
ED utilization rate | 6 months
  Rate of potentially avoidable emergency department utilization as determined by encounters recorded in health information exchange data and categorized using the NYU ED Algorithm.
Missed primary care appointments rate | 6 months
  Rate of no show / cancelled appointments at the intervention site primary care clinics as recorded in the intervention site's electronic health record system

SECONDARY OUTCOMES:
Hospitalization rate | 6 months
  Rate of all cause and potentially preventable hospitalization as determined by encounters recorded in health information exchange data and categorized using AHRQ's prevention quality indicator definitions

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R Vest, PhD, Principal Investigator — Associte Professor
Locations (1):
- Eskenazi Health, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kasthurirathne SN, Vest JR, Menachemi N, Halverson PK, Grannis SJ. Assessing the capacity of social determinants of health data to augment predictive models identifying patients in need of wraparound social services. J Am Med Inform Assoc. 2018 Jan 1;25(1):47-53. doi: 10.1093/jamia/ocx130. PMID 29177457
- [Background] Vest JR, Grannis SJ, Haut DP, Halverson PK, Menachemi N. Using structured and unstructured data to identify patients' need for services that address the social determinants of health. Int J Med Inform. 2017 Nov;107:101-106. doi: 10.1016/j.ijmedinf.2017.09.008. Epub 2017 Sep 20. PMID 29029685
- [Background] Vest JR, Menachemi N, Grannis SJ, Ferrell JL, Kasthurirathne SN, Zhang Y, Tong Y, Halverson PK. Impact of Risk Stratification on Referrals and Uptake of Wraparound Services That Address Social Determinants: A Stepped Wedged Trial. Am J Prev Med. 2019 Apr;56(4):e125-e133. doi: 10.1016/j.amepre.2018.11.009. Epub 2019 Feb 14. PMID 30772150